CLINICAL TRIAL: NCT04660877
Title: Anabolic Effects of Cheddar Cheese Consumption in Human Skeletal Muscle
Brief Title: Blood and Muscle Response to Cheddar Cheese in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Associate Professor, University of Utah
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 110963
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: Participants take part in an experiment in which they consume cheese then at another time consume milk
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cheddar chese (Experimental): Once enrolled, participants will either ingest 20 grams of protein from 1) cheese or 2) milk for the first Metabolic Study and then the other product when they return after the washout period (~1 month) for Metabolic Study #2.
  Interventions: Dietary Supplement: Cheddar Cheese
- Milk (Active Comparator): Once enrolled, participants will ingest 20 grams of protein from 1) cheese or 2) milk for the first Metabolic Study and then the other product when they return after the washout period (~1 month) for Metabolic Study #2.
  Interventions: Dietary Supplement: Milk

INTERVENTIONS:
Dietary Supplement: Cheddar Cheese — 20g of protein from cheddar cheese
  Arms: Cheddar chese
Dietary Supplement: Milk — 20g of protein from milk
  Arms: Milk

SUMMARY:
The goal of this project is to use a cross over design in young healthy male and female adults:

1. To determine the amino acid blood response to the acute ingestion of cheddar cheese in comparison to that of milk.
2. To determine the muscle mTORC1 response to the acute ingestion of cheddar cheese in comparison to that of milk.

DETAILED DESCRIPTION:
Each subject will take part in two metabolic studies. Each metabolic study was designed to test the acute blood and muscle response to an ingested amount of either cheddar cheese or milk. Approximately, one month after the first experiment (Metabolic Study #1), the participant will complete the second experiment (Metabolic Study #2) which was exact in design and at the same time of day as the first study but the participant ingested the alternate food product. The morning of the metabolic studies, the participant will arrive at the clinical research center after a 10h fast. A catheter will be placed in the participants' arm for blood sampling. Next, the participant will undergo a fasted thigh skeletal muscle biopsy. Following the muscle biopsy, the participant will consume either cheddar cheese (65g) or milk (370 mL) each amounting to 20g of protein. Subsequent muscle biopsies will occur at 60 and 180min after product ingestion. Blood sampling will occur in the fasted state and periodically after ingestion of the products (up to 300min).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35y

Exclusion Criteria:

1. History of cardiovascular disease
2. History of endocrine or metabolic disease (e.g., hypo/hyperthyroidism, diabetes)
3. History of kidney disease or failure
4. History of liver disease
5. History of respiratory disease (acute upper respiratory infection, chronic lung disease)
6. History of stroke with motor disability
7. Use of anticoagulant therapy (e.g., Coumadin, heparin) including aspirin and fish oils within 7d of the first biopsy experiment
8. Elevated systolic blood pressure >150 or a diastolic blood pressure > 100
9. Smoking
10. Recent anabolic or corticosteroids use (within 12 weeks)
11. Pregnancy as determined by a pregnancy test
12. self report of lactose intolerance
13. Any other medical condition or event considered exclusionary by the PI and faculty physician

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Response to cheese or milk ingestion | Area under the curve 0-300min after ingestion
  blood amino acids area under the curve in response to acute stimulation of cheese or milk consumption

SECONDARY OUTCOMES:
Response to cheese or milk ingestion | Change between 60min after ingestion and fasted response
  muscle mTORC1 change in response to acute stimulation of cheese or milk

CONTACTS AND LOCATIONS:
Overall Officials: Micah Drummond, Principal Investigator — University of Utah
Locations (1):
- The University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No